CLINICAL TRIAL: NCT05680116
Title: The Effect of Wearable Vibration Therapy on Shoulder Functionality in Individuals Receiving Adjuvant Radiotherapy After Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, Asistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATADEK 2022-17/27
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home based exercise group (Active Comparator): Patients who will start radiotherapy after breast cancer surgery will be evaluated prior to treatment. During the radiotherapy process, all of the patients will be included in the home exercise program, 5 days a week, 2 sessions a day, each exercise will be 10x2 repetitions. Exercise follow-up of the patients will be provided with weekly routine face-to-face checks. After an average of 6 weeks of radiotherapy, the initial evaluations will be repeated.
  Interventions: Other: Home based exercise
- Home based exercise plus vibration therapy group. (Experimental): Patients who will start radiotherapy after breast cancer surgery will be evaluated prior to treatment. During the radiotherapy process, all of the patients will be included in the home exercise program, 5 days a week, 2 sessions a day, each exercise will be 10x2 repetitions. The study group continues their home based exercise, in addition they will receive 30 minutes of Myovolt (Myovolt TM, Myovolt Limited, Christchurch, New Zealand) device which is wearable vibration therapy 2 days a week. The vibration program will continue for 6 weeks, in the form of 2 sessions per week. Intermittent and sinusoidal modes between 20-100 Hz will be used for the vibration frequency.
  Interventions: Device: MYOVOLT (MyovoltTM, Myovolt Limited, Christchurch, New Zealand ) wearable vibration therapy device

INTERVENTIONS:
Device: MYOVOLT (MyovoltTM, Myovolt Limited, Christchurch, New Zealand ) wearable vibration therapy device — Patients will wear Myovolt shoulder device twice a week and each session will continue 30minutes. This therapy will apply during the radiotherapy process. The device will be applied on the bare skin of the shoulder area. The first 10 minutes of the 30 minutes will be intermittent vibration, the other 20 minutes will be done in the sinusoidal vibration program. Both programs will be in the range of 20-100 Hz.
  Arms: Home based exercise plus vibration therapy group.
Other: Home based exercise — Patients will do home based exercise during the radiotherapy process. 5 days a week. 2 sessions a day, each exercise will be 10x2 repetitions
  Arms: Home based exercise group

SUMMARY:
The aim of our study is to investigate the effect of vibration therapy to be applied to patients undergoing breast cancer surgery and adjuvant radiotherapy on upper extremity joint range of motion, muscle strength, grip strength, pain, functionality, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer, undergoing breast-conserving surgery or having a total mastectomy and undergoing axillary lymph node dissection during surgery
* Cases that will start radiotherapy after surgery
* Being over 18 years old
* Absence of limitation in shoulder joint range of motion in preoperative evaluations.
* No speech and hearing problems
* Volunteering of the patients included in the study

Exclusion Criteria:

* Having previously undergone ipsilateral or contralateral breast cancer surgery
* Presence of active or metastatic cancer focus
* Presence of a neurological disease or orthopedic surgery affecting upper extremity functionality
* Carrying a pacemaker
* Presence of infection and open wound
* Finding a post-surgical drain
* Cases with mental and cooperation problems

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 6 weeks
  Hand-held dynamometer will be used to evaluate shoulder flexion, abduction, external and internal rotation muscles' strength
Range of motion | 6 weeks
  Shoulder range of motion will be evaluated by digital goniometer. Shoulder flexion degree, shoulder extension degree, abduction and adduction degree, internal rotation and external rotation degree will be assessed with digital goniometer. The results will be recorded in degrees.

SECONDARY OUTCOMES:
Pain - Visual Analogue Scale | 6 weeks
  Visual Analogue Scale is one of the simple and common methods used in pain assessment. Self reported pain intensity during the rest and the activity measured by 0-10 centimeter chart. Visual Analogue Scale (VAS), where 0 indicates no pain or best and 10 indicates the most intense pain imaginable or worst. The patient will mark the severity of the pain on a 10 cm long chart.
Grip strength | 6 weeks
  Grip strength was evaluated by hand grip dynamometry (Saehan Hydraulic Hand Dynamometer ) Measurements were performed in affected side according to positions defined by American Society of Hand Therapists (sitting with the shoulder adducted to the side and the elbow flexed 90° with the forearm and wrist in the neutral mid-position)
Disability | 6 weeks
  Disabilities of the Arm Shoulder and Hand ( DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms.The DASH questionnaire consists of three parts.The first part consists of 30 questions. 21 questions assess the difficulty of the patient in daily life activities, 5 question symptoms, and the remaining 4 questions assess social function, work, sleep, and self-confidence of the patient.In the DASH questionnaire, questions are answered in 5-point likert system. 1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not at all. The total score varies between 0 and 100 points and the low score indicates good health
Quality of Life- Functional Assessment of Cancer Therapy-Breast" (FACT-B) | 6 weeks
  It is designed to evaluate the quality of life in breast cancer patients from multiple perspectives. Its validity and reliability have been demonstrated. It consists of 5 subscales that assess quality of life as physical condition (7 questions), social life and family status (7 questions), emotional status (6 questions), activity status (7 questions), and other breast cancer-specific concerns (9 questions). The survey has 5-point likert scoring (0=not at all, 1=a little, 2=a little, 3=quite a lot, 4=a lot) . The total score is calculated by summing the subscale scores. A higher score on the questionnaire indicates a higher quality of life
Tone - Myoton® PRO | 6 weeks
  Myoton® PRO (Myoton Ltd, Myoton AS, Estonia) device will be used to objectively evaluate the measurement of Pectoralis Major muscle tone of the patients who will participate in the study. Myoton® PRO is a portable digital device that measures the tone with an objective and noninvasive method.
  A constant pre-pressure (0.18 N) is applied to the skin surface to compress the subcutaneous superficial tissues. The tension state of the tissue that characterized by the natural oscillation frequency; Hz.
Stiffness of Muscle- Myoton® PRO | 6 weeks
  Myoton® PRO (Myoton Ltd, Myoton AS, Estonia) device will be used to objectively evaluate the measurement of Pectoralis Major muscle stiffness of the patients who will participate in the study. Myoton® PRO is a portable digital device that measures the stiffness with an objective and noninvasive method.
  A constant pre-pressure (0.18 N) is applied to the skin surface to compress the subcutaneous superficial tissues. The stiffness of the tissue that characterized by the natural oscillation stiffness; N/m
Elasticity of Muscle -Myoton® PRO | 6 weeks
  Myoton® PRO (Myoton Ltd, Myoton AS, Estonia) device will be used to objectively evaluate the measurement of Pectoralis Major muscle elasticity of the patients who will participate in the study. Myoton® PRO is a portable digital device that measures the elasticity with an objective and noninvasive method.
  A constant pre-pressure (0.18 N) is applied to the skin surface to compress the subcutaneous superficial tissues. The elasticity of the tissue that characterized bythe logarithmic decrease of the natural oscillation;

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Feyzioğlu, PhD, Principal Investigator — Acibadem University
Locations (1):
- Professor Cemil Taşcıoğlu Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Feyzioglu O, Dincer S, Yilmaz BD, Saldiran TC, Ozturk O. Effects of Vibration Therapy on Muscle Strength, Shoulder Range of Motion, and Muscle Biomechanical Properties in Patients With Breast Cancer Undergoing Radiotherapy: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Apr 1;104(4):325-334. doi: 10.1097/PHM.0000000000002664. Epub 2024 Nov 14. PMID 39774038